CLINICAL TRIAL: NCT01517113
Title: Age-Associated Changes in Regional Adiposity and Novel Cardiovascular Risk Factors
Brief Title: Age-Related Changes in Body Composition
Status: Terminated | Type: Observational
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 120019; 12-AG-0019
Record Dates: First submitted 2012-01-24; First posted 2012-01-25 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2017-10-13

CONDITIONS: Hypertension; Atherosclerosis
Keywords: Endothelial Dysfunction; Hepatic; Adiposity; Cytokines; Muscle Mass; Coronary Artery Disease; Aging; Inflammation
MeSH Terms: conditions — Hypertension; Atherosclerosis; Obesity; Coronary Artery Disease; Inflammation

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- Advancing age is associated with greater risk of heart disease. High blood pressure and hardening of the arteries also have more complications with age. Studies suggest that age-related inflammation may affect fatty tissue in the body. If this fat develops in the muscles or around the heart, it may increase risks of heart disease. Researchers will study body composition in older adults to see if age-related changes in body fat are related to higher risks of heart disease.

Objectives:

- To study the relationship between fat deposits and aging, and greater risks of heart disease.

Eligibility:

* Participants in the Baltimore Longitudinal Study of Aging between 50 and 80 years of age.
* Individuals between 50 and 80 years of age who have been diagnosed with coronary artery disease.

Design:

* Participants will be screened with a physical exam and medical history.
* Participants will provide blood and urine samples. They will also have their height and weight measured. Waist circumference will also be taken.
* Participants will have a DEXA scan to study their muscles.
* Participants will have magnetic resonance imaging scans. These scans will study heart function and muscle and blood vessel health.
* Participants with coronary artery disease will have catheterization. Blood samples will be collected during the procedure....

DETAILED DESCRIPTION:
Advancing age is associated with an increasing prevalence, incidence, and complications of cardiovascular diseases, particularly hypertension and atherosclerosis. The reasons why age is associated with increased susceptibility to cardiovascular diseases are not understood but recent literature suggests that systemic inflammation, by affecting endothelial function, vascular stiffening, diastolic dysfunction and insulin resistance may be an important contributing cause. Aging is also associated with substantial changes in body composition, primarily an increase in fat mass and a decline in lean body mass. Studies in animal models and in humans have shown that the adipose tissue is an important source of pro-inflammatory mediators and suggested that changes in body composition may be the primary cause of the pro-inflammatory state of aging. A number of gene expression studies in animal models show that genes of several pro-inflammatory cytokines are over-expressed with aging, especially in the adipose tissue. The overproduction of pro-inflammatory cytokines have important systemic effects, including (1) endothelial dysfunction, one of the earliest features of atherosclerosis; (2) vascular stiffening, the primary etiology for isolated systolic hypertension in the elderly; and (3) insulin resistance, the principal metabolic abnormality associated with cardiovascular risk. Fat infiltration in the liver also promotes chronic inflammation both directly and by inducing apoptosis of hepatocytes with consequent inflammatory response and deterioration of liver function.

Limited data exists suggesting that deposition of adipose tissue in specific districts but not in others is associated with high circulating levels of pro-inflammatory markers. For example, in humans central adiposity, including fat accumulation surrounding the heart, and fat infiltration in the muscle, opposed to subcutaneous adiposity seems to be particularly pro-inflammatory. However, this information comes from small studies, or studies limited to a very narrow age-range. In addition, the assessment of regional adiposity was mostly based on anthropometrics. Indeed, non-invasive methodology for the assessment of regional lipid deposition profiles has become available only recently.

We propose to complement the BLSA population with a group of individuals with established CAD because the inclusion of this group may help to determine whether, and if so the extent to which, the expected relationships between body adiposity, inflammation, endothelial dysfunction, arterial stiffness and insulin resistance are different in healthy individuals compared to age-matched individuals with clinically overt vascular disease.

As a side hypothesis, we will also verify whether changes in Testosterone with age are associated with changes in regional fat accumulation. To test this hypothesis we will measure total, free and biovailable Testosterone in all participants.

ELIGIBILITY:
* INCLUSION CRITERIA: (both Group A and Group B):
* Age 50-90 years
* Body mass index greater than or equal to 20 and less than or equal to 35
* Weight is less than 300 lbs

In addition, for CAD participants (Group B):

* Catheterization-documented coronary artery disease, defined as greater than or equal to 70% stenosis in a major epicardial coronary artery, or greater than or equal to 50% stenosis of the left main coronary artery OR
* Prior myocardial infarction defined by ischemic symptoms associated with ECG changes and enzyme elevation.

In addition, for CAD participants in whom arterial and hepatic vein inflammatory mediators will be obtained:

- Scheduled for clinically indicated right or left heart catheterization, no contraindication for the procedure, and consented to the research procedure.

Exclusion criteria

* Known inflammatory disease
* Known liver disease
* Abnormal liver function tests defined by enzyme rise to greater than three times the upper limit of normal.
* Contraindications to the performance of MRI scans
* Chronic use of anti-inflammatory agents other than low dose aspirin (81mg). Chronic use is defined here as the inability to stop taking their anti-inflammatory agent for at least one week before starting this study
* Pregnant or lactating

In addition, for BLSA participants:

- Known coronary artery disease by prior history, examination, or resting or stress electrocardiogram testing.

In addition, for CAD participants undergoing arterial and hepatic vein inflammatory mediator sampling:

* Receiving therapy with heparin, a glycoprotein IIB/IIIA inhibitor, or bivalirudin
* History of atrial fibrillation
* Presence of an inferior vena cava filter
* Deep venous thrombosis
* Active infection.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-01-02; Study Completion 2017-10-13

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Ferrucci, M.D., Principal Investigator — National Institute on Aging (NIA)
Locations (2):
- United States (2):
  - Johns Hopkins University, Baltimore, Maryland
  - National Institute of Aging, Clinical Research Unit, Baltimore, Maryland

REFERENCES:
- [Background] Singh T, Newman AB. Inflammatory markers in population studies of aging. Ageing Res Rev. 2011 Jul;10(3):319-29. doi: 10.1016/j.arr.2010.11.002. Epub 2010 Dec 8. PMID 21145432
- [Background] Ferrucci L, Corsi A, Lauretani F, Bandinelli S, Bartali B, Taub DD, Guralnik JM, Longo DL. The origins of age-related proinflammatory state. Blood. 2005 Mar 15;105(6):2294-9. doi: 10.1182/blood-2004-07-2599. Epub 2004 Nov 30. PMID 15572589
- [Background] Brooks GC, Blaha MJ, Blumenthal RS. Relation of C-reactive protein to abdominal adiposity. Am J Cardiol. 2010 Jul 1;106(1):56-61. doi: 10.1016/j.amjcard.2010.02.017. Epub 2010 May 13. PMID 20609648